CLINICAL TRIAL: NCT02629224
Title: Pharmacokinetic (PK) Study of ASP8825 - Evaluation of Pharmacokinetics in Patients With Impaired Renal Function and Haemodialysis
Brief Title: ASP8825 - Pharmacokinetics Study in Patients With Impaired Renal Function and Haemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8825-CL-0012
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Patients With Impaired Renal Function and Haemodialysis
Keywords: Impaired renal function; Haemodialysis; ASP8825; XP13512
MeSH Terms: conditions — Renal Insufficiency | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal impairment (Experimental)
  Interventions: Drug: ASP8825
- Haemodialysis (Experimental)
  Interventions: Drug: ASP8825

INTERVENTIONS:
Drug: ASP8825 — Oral
  Other Names: gabapentin enacarbil

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics and safety of ASP8825 in patients with impaired renal function and haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: ≥40.0 kg and <80.0 kg
* Body mass index BMI: ≥16.0 and <30.0 [BMI= Body weight (kg)/(Height (m))2]
* For Renal impairment patients: Patients with eGFR by GFR predictive equation for Japanese within < 50 mL.min/1.73m2 at screening and who is not undergoing dialysis
* For Haemodialysis patients: Patients who receive dialysis at screening
* Patients whose treatment regimen (including diet) for renal impairment or complications remain unchanged within 14 days prior to dosing, or patients who receive treatments (including diet) that need not to be changed during the period from 14 days before dosing to follow-up examination in the opinion of the investigator or sub-investigator.
* Female subjects who agree use effective contraception starting at informed consent and throughout the study period

Exclusion Criteria:

* Patients with a complication or history of the inappropriate for this study (except for a complication of primary disease for renal dysfunction, like diabetes etc., or complication of hypertension or anemia etc.)
* Patients with a complication or history of recurring alimentary disease
* Patients with a history of gastrointestinal surgical operation
* Patients with a complication of severe heart disease
* Patients with a complication or history of malignant tumor (However, a patient without recurrence of the malignant tumor for more than 5 years after the treatment may be eligible for the study.)
* Patients judged ineligible by the investigator or sub-investigator based on the results of medical examination, vital sign, 12-ECG and laboratory test
* Patients who have an Hb value <9g/dL at screening
* Patients who received or are scheduled to receive any study drugs in other clinical trials or post-marketing studies within 120 days before screening
* Patients who received or are scheduled to receive medications within seven days before the dosing of the investigational drug
* Patients who previously received administration of Gabapentin or ASP8825

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of gabapentin in plasma: Cmax in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  Cmax: Maximum concentration
PK parameters of gabapentin in plasma: tmax in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  tmax: Time of Cmax
PK parameter of gabapentin in plasma: AUC24h in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  AUC24h: Area under the concentration-time curve from the time of dosing to 24hours after dosing
PK parameter of gabapentin in plasma: Cmax in Haemodialysis patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 25, 26, 27, 28, 30, 36 and 48 hr after dosing
  Cmax: Maximum concentration
PK parameters of gabapentin in plasma: tmax in Haemodialysis patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 25, 26, 27, 28, 30, 36 and 48 hr after dosing
  tmax: Time of Cmax
PK parameter of gabapentin in plasma: AUC24h in Haemodialysis patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 25, 26, 27, 28, 30, 36 and 48 hr after dosing
  AUC24h: Area under the concentration-time curve from the time of dosing to 24hours after dosing
PK parameters of gabapentin in plasma: AUClast in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  AUClast: Area under the concentration-time curve from the time of dosing to the last measurable concentration
PK parameter of gabapentin in plasma: AUCinf in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameters of gabapentin in plasma: kel in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  kel: Elimination rate constant
PK parameters of gabapentin in plasma: t1/2 in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  t1/2: Terminal elimination half-life
PK parameters of gabapentin in plasma: CL/F in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  CL/F: Apparent total systemic clearance
PK parameters of gabapentin in plasma: Vz/F in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  Vz/F: Apparent volume of distribution during the terminal elimination phase
PK parameters of gabapentin in plasma: MRTinf in Renal impairment patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hr after dosing
  MRTinf: Mean residence time from the time of dosing extrapolated to time infinity
PK parameters of gabapentin in plasma: t1/2, pre in Haemodialysis patients | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 18 hr after dosing
  t1/2, pre: Elimination half-life for pre-hemodialysis
PK parameters of gabapentin in plasma: t1/2, HD in Haemodialysis patients | 24, 25, 26, 27 and 28 hr after dosing
  t1/2,HD: Elimination half-life for hemodialysis
PK parameters of gabapentin in plasma: t1/2, post in Haemodialysis patients | 30, 36 and 48 hr after dosing
  t1/2, post: Elimination half-life for post-hemodialysis
PK parameters of gabapentin: CLDP in Haemodialysis patients | 25, 26, 27 and 28 hr after dosing
  CLDP: Hemodialysis clearance calculated from the concentration of gabapentin at pre-dialyzer and post-dialyzer
PK parameters of gabapentin in plasma: AUCD in Haemodialysis patients | 24, 25, 26, 27 and 28 hr after dosing
  AUCD: Area under the concentration-time curve from the start to end of haemodialysis the concentration of gabapentin in plasma pre-dialyzer
PK parameters of gabapentin in urine: Ae72h in Renal impairment patients | Up to 72 hr after dosing
  Ae72h: Amount of gabapentin excreted into the urine from the time of dosing to 72 hr after dosing
PK parameters of gabapentin in urine: Ae%72h in Renal impairment patients | Up to 72 hr after dosing
  Ae%72h: Percent of gabapentin excreted into the urine from the time of dosing to 72 hr after dosing
PK parameters of gabapentin in urine: CLR in Renal impairment patients | Up to 72 hr after dosing
  CLR: Renal clearance
PK parameters of gabapentin in urine: Ae48h in Haemodialysis patients | Up to 48 hr after dosing
  Ae48h: Amount of gabapentin excreted into the urine from the time of dosing to 48 hr after dosing
PK parameters of gabapentin in urine: Ae%48h in Haemodialysis patients | Up to 48 hr after dosing
  Ae%48h: Percent of gabapentin excreted into the urine from the time of dosing to 48 hr after dosing
PK parameters of gabapentin in dialyzing fluid: Adt in Haemodialysis patients | Up to 48 hr after dosing
  Adt: Cumulative amount in dialyzing fluid from the time of dosing to time after dosing
PK parameters of gabapentin in dialyzing fluid: Adt% in Haemodialysis patients | Up to 48 hr after dosing
  Adt%: Excretion rate in dialyzing fluid
PK parameters of gabapentin in dialyzing fluid: CLDD in Haemodialysis patients | Up to 48 hr after dosing
  CLDD: Hemodialysis clearance calculated from the Cumulative amount in dialyzing fluid
Safety assessed by AEs | Up to 7 days after the study drug dosing
  AEs: Adverse Events
Safety assessed by Vital signs | Up to 7 days after the study drug dosing
  Supine blood pressure, supine pulse rate and axillary body temperature
Safety assessed by Laboratory tests | Up to 7 days after the study drug dosing
  Hematology, blood biochemistry, and urinalysis
Safety assessed by 12-lead ECGs | Up to 7 days after the study drug dosing
  ECG: Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Fukuoka
  - Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=8825-CL-0012